CLINICAL TRIAL: NCT04691011
Title: New Magnetic Resonance Imaging Biomarkers in Amyotrophic Lateral Sclerosis
Acronym: IRM-SLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-50
Record Dates: First submitted 2020-10-22; First posted 2020-12-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: 3 groups :
  * muscle
  * brain
  * spinal cord
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle (Other)
  Interventions: Other: Muscular MRI; Other: Electrophysiological exam
- Spinal cord (Other)
  Interventions: Other: Muscular MRI; Other: Electrophysiological exam; Other: Spinal cord MRI
- Brain (Other)
  Interventions: Other: Muscular MRI; Other: Electrophysiological exam; Other: Brain MRI

INTERVENTIONS:
Other: Muscular MRI — MRI (1.5T)
Other: Electrophysiological exam — MUNIX
Other: Brain MRI — MRI (7T)
  Arms: Brain
Other: Spinal cord MRI — 7T and 3T MRI
  Arms: Spinal cord

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disabling and rapidly progressive neurodegenerative disorder. There is no treatment that significantly slows progression. Our project aims to find new biomarkers in MRI at three levels: cerebral, medullary and muscular. These markers could allow an earlier diagnosis of the disease by showing more specific lesions of ALS and to quantify these lesions to measure the progression of the disease. This study will use advanced Magnetic Resonance Imaging (MRI) techniques High field (3T) and very high field (7T) MRI. Results from neurological and electrophysiological tests will be compared to the MRI. Subjects will be recruited from ALS center of Marseille, France. MRI will be done on ALS patients at baseline, at 3 month and at 6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be adults with a diagnosis of ALS.
* Healthy controls will also be recruited and will be age- and gender-matched to patients.
* Patients able to undergo a brain MRI for approximately an hour.

Exclusion Criteria:

* Subjects with other psychiatric or CNS or PNS diseases.
* Subjects ineligible for MRI investigation due to a pacemaker or other metallic foreign body, or significant claustrophobia that could affect the ability to have an MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Disease progression using MRI | Change from Baseline and at Month 6
  Muscular, brain and spinal cord MRI (brain sodium concentration, muscular volume of members, measure of transversal area for spinal cord)

SECONDARY OUTCOMES:
Link between MRI and clinical scales | Baseline and Month 6
  ALSFRS score, MRC score, ECAS score
Link between MRI and MUNIX | Baseline and Month 6
  For muscle, brain and spinal cord group
Alterations of metabolic and funtional brain | Baseline and Month 6
  Multiparametric MRI (diffusion parameters, myelin parameters, quantification of fat-infiltration and oedema)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido Pradalié, Study Director — Direction Recherche Santé APHM
Locations (1):
- Shahram Attarian, Marseille, France